CLINICAL TRIAL: NCT00613821
Title: A Comparison of Intrauterine Lidocaine Infusion and Paracervical Block for Pain Management in First Trimester Abortions
Brief Title: Lidocaine and Pain Management in First Trimester Abortions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Alison Edelman, Assistant Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OHSU RES 2173
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Results first posted 2017-07-31 (Actual); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Pain
Keywords: surgical abortion; pain management
MeSH Terms: conditions — Pain; Agnosia | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine infusion (Experimental): 5 milliliter intrauterine infusion of 4% lidocaine, infusion will be placed slowly over 3 minutes.
  Interventions: Drug: Lidocaine
- Paracervical block only (Active Comparator): Standard paracervical block (8 milliliter 1% lidocaine at 4 and 8 o'clock at the cervical-vaginal reflection) will be placed.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — 5 milliliter intrauterine infusion of 4% lidocaine, infusion will be placed slowly over 3 minutes.
  Arms: Lidocaine infusion
Drug: Lidocaine — Standard paracervical block (8 milliliter 1% lidocaine at 4 and 8 o'clock at the cervical-vaginal reflection) will be placed.
  Arms: Paracervical block only

SUMMARY:
The purpose of this study is to examine the effect of lidocaine (a numbing medication) inside the uterus on patient pain during an early abortion, compared to the paracervical block (lidocaine injected on either side of the cervix).

DETAILED DESCRIPTION:
The Investigators intend to conduct a randomized, patient-blinded control trial at Oregon Health and Science University and Planned Parenthood of the Columbia Willamette. Women will be approached about this study after they have made a decision to terminate the pregnancy. The women will be blinded and randomized into one of two study arms.

Group 1: the investigator will apply pressure with the capped needle of the paracervical block at the cervical-vaginal reflexion at 4 and 8 o'clock. This will approximate the steps involved in a paracervical block without injecting the patient. Following this, the patient will receive a 5 milliliter intrauterine infusion of 4% lidocaine using a sterile 3mm Novak curette. The infusion will be placed slowly over 3 minutes.

Group 2: a standard paracervical block (8 milliliter 1% lidocaine at 4 and 8 o'clock at the cervical-vaginal reflection) will be placed. Following this, a 3 mm Novak curette will be placed in the vagina and held to the external os of the cervix for 3 minutes. The curette will not be placed through the cervix and no infusion will be performed. This will approximate the steps involved in an intrauterine infusion without injecting the patient.

During the procedure, women in both groups will be asked to rate their pain at various times using a 10 cm visual analog scale (VAS).

ELIGIBILITY:
Inclusion Criteria:

* Good general health
* Age>18years
* English speaking
* Voluntarily requesting pregnancy termination
* Have an estimated gestation of up to 76 days since the first day of the preceding menstrual period
* Confirmed by ultrasound
* Be able and willing to sign an informed consent
* Agree to the terms of the study
* All patients must be premedicated with Ibuprofen and Valium (per clinic protocols)

Exclusion Criteria:

* Significant physical or mental health condition
* A gestational age of 77 days or more
* Adnexal mass or tenderness on pelvic exam consistent with pelvic inflammatory disease
* Patients who require or request IV/intramuscular sedation
* Patients who refuse Ibuprofen, Valium and/or paracervical blocks
* Patients allergic to lidocaine
* Patients with known hepatic disease
* Patients weighing less than 100 lbs

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2007-09; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alison Edelman, M.D., M.P.H, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Planned Parenthood of the Columbia Willamette, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon

REFERENCES:
- [Background] Edelman A, Nichols MD, Leclair C, Jensen JT. Four percent intrauterine lidocaine infusion for pain management in first-trimester abortions. Obstet Gynecol. 2006 Feb;107(2 Pt 1):269-75. doi: 10.1097/01.AOG.0000194204.71925.4a. PMID 16449111

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lidocaine Infusion | Paracervical Block Only
Started | 40 | 40
Completed | 38 | 39
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lidocaine Infusion | Paracervical Block Only | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 40 | 80
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: The Effects of an Intrauterine Lidocaine Infusion to Standard Paracervical Block on Decreasing Patient Pain Measured by Visual Analog Scale in First Trimester Abortions.
Description: Subjects perception of pain is measured using a 100mm visual analog scale (VAS).The 100mm Pain Visual Analog Scale (VAS) is an instrument used to capture subjective attitudes that cannot be directly measured. When responding to a VAS item, respondents specify their level of pain by indicating a position along a 100mm continues line: pain scores can range from 0 (no pain) to 100 (worst pain imaginable).
Time Frame: Immediately (time zero) at uterine aspiration
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Lidocaine Infusion | Paracervical Block Only
Number analyzed (Participants) | 40 | 40
mm | 71 (20) | 43 (30)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected at procedure visit and follow up visit, 2 weeks post-procedure.
Arm/Group | Lidocaine Infusion | Paracervical Block Only
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/40
Other Adverse Events (participants affected / at risk) | 1/40 | 3/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lidocaine Infusion (N=40) | Paracervical Block Only (N=40)
Immediate reaspiration (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Needed antibiotics at follow up visit (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Delayed reaspiration (Reproductive system and breast disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No